CLINICAL TRIAL: NCT01191411
Title: Increasing Colorectal Cancer Screening in a Safety-net Health System With a Focus on the Uninsured: Benefits and Costs.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other); Polymedco Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: STU 012011-152
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal neoplasms; screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mailed invitations for FIT test kits (Active Comparator): Fecal Immunochemical Tests (FIT) kits from Polymedco Incorporated are mailed to patients' homes for free colorectal cancer screening.
  Intervention: Screening for colorectal cancer using a Polymedco home FIT kit. Mailed invitation to complete a free one sample home FIT kit. Automated and live phone call reminders to promote screening completion, plus usual medical care.
  Patients with abnormal FIT results are navigated to complete a diagnostic colonoscopy.
  Interventions: Other: Mailed invitations for FIT test kits
- Mailed invitations for a colonoscopy (Active Comparator): Invitation to schedule a colonoscopy are mailed to patients' homes for free colorectal cancer screening.
  Intervention: Screening for colorectal cancer with colonoscopy. Mailed invitation to complete one free colonoscopy. Automated and live phone reminders to promote screening completion, plus usual medical care.
  Patients with abnormal polyps or adenomas will follow standard clinical protocol after their procedure.
  Interventions: Other: Mailed invitations for a colonoscopy
- Visit Based Care (Active Comparator): No invitation to complete colorectal cancer screening.
  Intervention: Usual medical care. Patients will continue to see their regular physician, and follow their physician's regular standard of care.
  Interventions: Other: Visit Based Care

INTERVENTIONS:
Other: Mailed invitations for FIT test kits — Mailed invitations for the non-invasive immunochemical stool blood test will be the intervention compared to the standard care at John Peter Smith Hospital. Patients will be invited to complete a free home-based, non-invasive immunochemical stool blood test.
  Other Names: Polymedco Fecal Immunochemical Test
  Arms: Mailed invitations for FIT test kits
Other: Mailed invitations for a colonoscopy — These patients will be mailed invitations to directly book a free colonoscopy, or to see a physician for free pre-operative screening at John Peter Smith Hospital.
  Arms: Mailed invitations for a colonoscopy
Other: Visit Based Care — Visit based standard care at John Peter Smith Hospital. Patients will continue to see their regular physician and follow the physician's recommendations as they normally would.
  Arms: Visit Based Care

SUMMARY:
Colon cancer (CRC) is a leading cause of cancer death in the United States. Screening can prevent CRC death, but screening rates are suboptimal, especially for vulnerable populations such as those with limited or no health insurance. This striking public health challenge demands urgent implementation of evidence-based strategies to reduce avoidable CRC death.

Prior research has shown that a direct-to-consumer strategy of inviting patients by mail to complete CRC screening may result in increased rates of screening completion. However, this approach has not been tested extensively in vulnerable populations, such as the under/uninsured, and minority populations often cared for by safety-net health systems. Further, it is unclear whether patients are more likely to participate in one CRC screening test versus another. Knowing this is important to designing programs for increasing screening. For example, the planning and resources required for a screening program with colonoscopy--which is a sensitive but invasive and expensive test--are very different from a program with that uses stool testing to detect microscopic blood such as an immunochemical stool blood test--which is a less sensitive, but non-invasive and cheap test.

Also, it is possible designing a program with a less sensitive, but more acceptable test could prevent more CRC death if participation in screening is test specific. For example, if many more patients participate in an immunochemical stool blood test based program than a colonoscopy based program, even though the immunochemical stool blood test is less sensitive, the program may save more lives because more patients are reached.

The aims of this trial are to:

Aim 1. Deliver CRC screening services (mailed invitation to screening, telephone reminders, and systematic clinical follow up) to uninsured, unscreened patients cared for by the safety-net health system serving Tarrant County, Texas. Patients will be invited to either:

1. Complete a free home-based, non-invasive immunochemical stool blood test
2. Complete a free colonoscopy

Aim 2. Evaluate program outcomes, including screening rates, cancers detected, and program costs.

The primary outcome is screening completion.

DETAILED DESCRIPTION:
Program setting. The John Peter Smith Hospital Health System (JPS) is a safety-net health care system serving Tarrant County, Texas (including Fort Worth), with over 850,000 yearly patient encounters. JPS qualifies as a safety-net health system based on a commitment to deliver health care to uninsured, Medicaid participants, and other vulnerable patients18, and is recognized as a disproportionate share hospital. JPS offers a tax-subsidized charity medical program called JPS Connection for uninsured Tarrant County residents who are not eligible for state or federal assistance programs such as Medicaid, with qualification based on federal poverty income levels.

Target population. Our specific project target population includes men and women, aged 54 to 64, without prior CRC screening, of all races/ethnicities (including African Americans, Hispanics, and Whites), who are primary English or Spanish language speaking, and uninsured but enrolled in the JPS Connection medical assistance program. We include only those individuals who qualify and are enrolled in the JPS Connection medical assistance program to ensure that all included patients have access to a primary provider, as well as surgical and medical cancer care, in the event that a patient has a cancer diagnosed.

TREATMENT (INTERVENTION) We will screen the administrative dataset that we are using to identify potential study participants for individuals who meet inclusion criteria. All patients selected to one of the programmatic screening approaches (Mailed FIT or Mailed Colonoscopy invitation) will receive the same, structured approach for encouragement of completion of CRC screening with the exception of the initial screening modality offered (e.g. FIT or colonoscopy). In addition, patients selected for program intervention will also be free to engage in usual medical care, and any associated visit-based screening at the discretion and preference of the individual and primary medical provider.

Mailed invitation program procedures. Every 3 months, ¼ of the patient group selected for the mail out program will receive an electronic, automated phone call, alerting them that an invitation to participate in CRC screening will be mailed to them shortly. All invitees, regardless of screen-group, will receive: 1) Invitation to participate in CRC screening with a specific test, including discussion of importance of screening, 2) Return card that may request to not participate in screening/be contacted in the future ("opt out" request). The invitations will be sent every 3 months in batches, rather than all at once, to allocate manpower resources for program follow up, and colonoscopy services as necessary for positive tests or screening requests.

Alert and reminder phone calls. At time of initial mailing of the invitation, a "TeleVox©" automated phone message, with a pre-recorded script (in both English and Spanish) will be generated to alert participants that an invitation is "in-the-mail." Fourteen days after initial mailing of the invitation, a "TeleVox©" automated reminder to respond to the invitation for screening with a pre-recorded script (in both English and Spanish) will be generated for all participants. Twenty-one to 36 days after initial invitation to testing, a "live" reminder phone call will be initiated by the screening coordination team for all individuals who have not responded to screening invitation. Up to 2 attempts will be made to contact individuals via phone; reaching a voice mail, an adult household member, or the target study participant will be considered a successful attempt. Reaching a disconnected, busy line, or line that rings with no answer on two attempts will be considered unsuccessful attempt. Continued intervention and follow up will not be based on whether or not phone call attempts were successful-all patients included in the program will be assessed for the outcome of screening participation.

Invitation letters. The invitation letters for screening with FIT or colonoscopy will contain the following elements: 1) Statement that risk of getting colon cancer increases with age and that screening can reduce the consequences, 2) Invitation to a specific modality, (FIT or colonoscopy) with a succinct description of the test, 3) Number to call with questions, 4) In the case of colonoscopy invitation, number to call to sign up, 5) Signature from a physician at JPS.

FIT procedures. Individuals assigned to FIT will be provided with written instructions on how to collect the stool samples for FIT testing. Kits will be mailed using return envelopes with pre-paid postage to a JPS.

Colonoscopy procedures. The colonoscopy invitation will consist of an explanation of colonoscopy, as well as a phone number to call to schedule a colonoscopy ("direct book") or a pre-colonoscopy clinic visit. The decision to "direct book" for colonoscopy or to arrange for a pre-colonoscopy clinic visit will be based on screening nurse phone interview using a short screening form. If potential medical contraindications to colonoscopy are noted, a pre-colonoscopy visit will be scheduled with a physician at JPS. Patients with uncontrolled medical conditions will be referred to primary physicians for further management and to consider CRC screening once the condition is under control. Reasons for not scheduling colonoscopy will be documented. The patient will receive a date and time assignment for the colonoscopy procedure, and instructions on bowel preparation for the procedure. The preparation kit will be mailed to the patient's home. Reminder calls 5-7 days prior to the procedure to confirm the date and time of the procedure, review bowel preparation instructions, and answer any questions will occur. The day of the procedure, a history and physical will be performed to re-assess for any contraindications for colonoscopy. Polyps identified will be removed completely, with repeat colonoscopy and/or surgery if polyp removal not successful. Any mass lesions and any areas of inflamed or irregular colon mucosa will undergo biopsy. Endoscopy findings will be reviewed with each participant.

Test Follow Up. Individuals with positive FIT will be contacted to schedule a colonoscopy, with the goal of test completion within 8-12 weeks of test positivity. If phone contact for test scheduling cannot be established, a certified letter will be sent. Individuals with findings of adenoma or cancer on colonoscopy will be scheduled for a follow up, post-colonoscopy visit with the endoscopist who performed the procedure. Individuals with normal FIT or colonoscopy screening tests will have a letter mailed to his or her home, as well as the primary outpatient clinic identified by administrative data.

ELIGIBILITY:
Inclusion Criteria:

* 54 to 64 year old men and women
* All races and ethnicities
* Patients that have been on JPS Connection in 2010 or JPS Connection in 2009 and have been seen at least once between September 1, 2009 and August 31, 2010 in any JPS setting

Exclusion Criteria:

* No address and phone number on file
* Incarcerated individuals
* Primary language other than English or Spanish
* Up to date with CRC screening, defined as any:

  1. Fecal Occult Blood Test (FOBT) in 2009
  2. Flexible Sigmoidoscopy 2005-09
  3. Barium Enema 2005-09
  4. Colonoscopy 2002-09* Prior history of CRC, inflammatory bowel disease, or colorectal polyps.

Ages: 54 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5970 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith E Argenbright, MD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta S, Halm EA, Rockey DC, Hammons M, Koch M, Carter E, Valdez L, Tong L, Ahn C, Kashner M, Argenbright K, Tiro J, Geng Z, Pruitt S, Skinner CS. Comparative effectiveness of fecal immunochemical test outreach, colonoscopy outreach, and usual care for boosting colorectal cancer screening among the underserved: a randomized clinical trial. JAMA Intern Med. 2013 Oct 14;173(18):1725-32. doi: 10.1001/jamainternmed.2013.9294. PMID 23921906

RESULTS

PARTICIPANT FLOW:
Groups:
- Mailed Invitations for FIT Test Kits: Fecal Immunochemical Tests (FIT) kits from Polymedco Incorporated are mailed to patients' homes for free colorectal cancer screening.
  Intervention: Screening for colorectal cancer using a Polymedco home FIT kit. Mailed invitation to complete a free one sample home FIT kit. Automated and live phone call reminders to promote screening completion, plus usual medical care.
  Patients with abnormal FIT results are navigated to complete a diagnostic colonoscopy.
  Mailed invitations for FIT test kits: Mailed invitations for the non-invasive immunochemical stool blood test will be the intervention compared to the standard care at John Peter Smith Hospital. Patients will be invited to complete a free home-based, non-invasive immunochemical stool blood test.
- Mailed Invitations for a Colonoscopy: Invitation to schedule a colonoscopy are mailed to patients' homes for free colorectal cancer screening.
  Intervention: Screening for colorectal cancer with colonoscopy. Mailed invitation to complete one free colonoscopy. Automated and live phone reminders to promote screening completion, plus usual medical care.
  Patients with abnormal polyps or adenomas will follow standard clinical protocol after their procedure.
  Mailed invitations for a colonoscopy: These patients will be mailed invitations to directly book a free colonoscopy, or to see a physician for free pre-operative screening at John Peter Smith Hospital.
- Visit Based Care: No invitation to complete colorectal cancer screening.
  Intervention: Usual medical care. Patients will continue to see their regular physician, and follow their physician's regular standard of care.
  Visit Based Care: Visit based standard care at John Peter Smith Hospital. Patients will continue to see their regular physician and follow the physician's recommendations as they normally would.
Period: Overall Study
Arm/Group | Mailed Invitations for FIT Test Kits | Mailed Invitations for a Colonoscopy | Visit Based Care
Started | 1593 | 479 | 3898
Completed | 648 | 118 | 471
Not Completed | 945 | 361 | 3427

BASELINE CHARACTERISTICS:
Population: Men and women, aged 54 to 64 years, who were uninsured but enrolled in the JPS medical assistance program for the uninsured. Not up-to-date with colorectal cancer screening; no history of colorectal cancer, inflammatory bowel disease, or colorectal polyps.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mailed Invitations for FIT Test Kits | Mailed Invitations for a Colonoscopy | Visit Based Care | Total
Number analyzed (Participants) | 1593 | 479 | 3898 | 5970
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (3) | 59 (3) | 59 (3) | 59 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 993 | 286 | 2517 | 3796
  Male | 600 | 193 | 1381 | 2174
Race/Ethnicity, Customized [Number; unit: participants]
  White | 653 | 195 | 1600 | 2448
  Black | 370 | 128 | 913 | 1411
  Hispanic | 445 | 122 | 1140 | 1707
  Other | 125 | 34 | 245 | 404
Primary Language [Number; unit: participants]
  English | 1322 | 410 | 3253 | 4985
  Spanish | 271 | 69 | 645 | 985

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Cancer Screening Participation, Defined as Completion of a Guaiac or Immunochemical Stool Occult Blood Test, Colonoscopy, Sigmoidoscopy, or Barium Enem.
Description: To compare participation rates for screening between those receiving (a) mailed invitation to screening (immunochemical stool blood test (MailFIT) or colonoscopy(MailColo)) and (b) traditional visit-based screening (VisitBased), rates for these groups will be contrasted via a Chi-squared test. A p value<0.025 will be considered statistically significant.
Time Frame: 1 year
Population: Overall, out of 1593 patients assigned to FIT outreach, 648 were screened; out of 479 assigned to colonoscopy outreach, 118 were screened; and out of 3898 assigned to usual care, 471 were screened.
Measure: Number; unit: percentage of participants
Groups:
- Mailed Invitations for FIT Test Kits: Fecal Immunochemical Tests (FIT) kits from Polymedco are mailed to patients' homes for free colorectal cancer screening.
  Intervention: Screening for colorectal cancer using a Polymedco home FIT kit. Mailed invitation to complete a free one sample home FIT kit. Automated and live phone call reminders to promote screening completion, plus usual medical care.
  Patients with abnormal FIT results are navigated to complete a diagnostic colonoscopy.
  Mailed invitations for FIT test kits: Mailed invitations for the non-invasive immunochemical stool blood test will be the intervention compared to the standard care at John Peter Smith Hospital. Patients will be invited to complete a free home-based, non-invasive immunochemical stool blood test.
Arm/Group | Mailed Invitations for FIT Test Kits | Mailed Invitations for a Colonoscopy | Visit Based Care
Number analyzed (Participants) | 1593 | 479 | 3898
percentage of participants
  All groups - screened | 40.7 | 24.6 | 12.1
  Men - screened | 38.7 | 23.3 | 10.7
  Women - screened | 41.9 | 25.2 | 12.8
  Whites - screened | 34.2 | 20.5 | 9.4
  Blacks - screened | 43 | 26.6 | 15.2
  Hispanics - screened | 48.1 | 28.7 | 13.2
  Other races/ethnicities - screened | 41.6 | 26.5 | 12.7

ADVERSE EVENTS:
Time Frame: Data for reporting serious adverse event was collected over a 3 month period.
Arm/Group | Mailed Invitations for FIT Test Kits | Mailed Invitations for a Colonoscopy | Visit Based Care
Serious Adverse Events (participants affected / at risk) | 1/1593 | 0/479 | 0/3898
Other Adverse Events (participants affected / at risk) | 0/1593 | 0/479 | 0/3898
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Mailed Invitations for FIT Test Kits (N=1593) | Mailed Invitations for a Colonoscopy (N=479) | Visit Based Care (N=3898)
Serious Adverse Event - Perforated cecum (Injury, poisoning and procedural complications) | 1/1 (1) | 0/0 (0) | 0/0 (0) — Routine colonoscopy scheduled prior to abnormal FIT results. Colonoscopy complication resulted in perforated cecum. Subject received surgical correction. Serious adverse event assessed as non-study related as procedure was part of usual medical care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No